CLINICAL TRIAL: NCT03588117
Title: Impact of Physician-supervised Nonsurgical Weight Management Program on Metabolic Syndrome
Brief Title: Prospective Metabolic Indicator Study
Acronym: PROMIS
Status: Completed | Type: Observational
Sponsor: Medi-Weightloss Franchising USA, LLC (Industry)
Responsible Party: Principal Investigator, Macklin E. Guzmán, Chief Science Officer, Medi-Weightloss Franchising USA, LLC
Other Study IDs: MWLCT01
Record Dates: First submitted 2018-05-10; First posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants of a weight management program: Participants of a physician-supervised nonsurgical weight management program were observed as they received weekly in-person coaching sessions with licensed clinicians. In-person coaching sessions were focused on educating participants on strategies to manage their weight and adopt a healthy lifestyle. Prescribed diets were individualized based on each participant's behavior, level of physical activity, and total energy expenditure. Supplements, appetite suppressant medications, and compounded injections were used to control appetite and/or boost energy during a period of low-caloric intake. The program was generally divided into three phases: Acute, Short-Term Maintenance, and Wellness.
  Interventions: Behavioral: Physician-supervised nonsurgical weight management program

INTERVENTIONS:
Behavioral: Physician-supervised nonsurgical weight management program — Participants of a physician-supervised nonsurgical weight management program were observed as they received weekly in-person coaching sessions with licensed clinicians. In-person coaching sessions were focused on educating participants on strategies to manage their weight and adopt a healthy lifestyle. Prescribed diets were individualized based on each participant's behavior, level of physical activity, and total energy expenditure. Supplements, appetite suppressant medications, and compounded injections were used to control appetite and/or boost energy during a period of low-caloric intake. The program was generally divided into three phases: Acute, Short-Term Maintenance, and Wellness.

SUMMARY:
The aim of this study was to assess the impact of a physician-supervised non-surgical medical weight management program on prevalence of metabolic syndrome and to examine the relationship between program retention and levels of key indicators of metabolic syndrome among participants that self-enrolled to the program. A total of 479 overweight or obese participants aged 19 years or older were observed. The revised National Cholesterol Education Program Adult Treatment Panel III (NCEP ATP III) criteria were used to define metabolic syndrome.

DETAILED DESCRIPTION:
Each individual self-enrolled to a physician-supervised non-surgical weight management program, hereafter referred to as the Program. They received a weight loss intervention as a part of routine medical care in the Program. At the end of their first consultation, each individual that met the inclusion criteria and failed to meet the exclusion criteria was asked if he or she would like to join the study. Each individual was informed that the study would not change the type or level of care that he or she would receive while enrolled to the program; however, researchers would be studying the effects of their care through additional screenings. Individuals who thereafter signed an informed consent form were monitored for changes in health outcomes without change to the Program.

This study was observational. Health outcomes were assessed in individuals that predefined their program status (i.e., enrolled or not enrolled). Each participant received routine medical care, and the investigators studied the effects of the intervention. No new intervention or intervention specific to participants only was assigned.

ELIGIBILITY:
Inclusion Criteria:

* The patient is at least 18 years of age.
* The patient is overweight or obese (BMI≥25 kg/m2).

Exclusion Criteria:

- The patient was previously enrolled in the Medi-Weightloss program

Ages: 19 Years to 83 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: New patients of the Medi-Weightloss franchise, a physician-supervised nonsurgical weight management program
Sampling Method: Non-Probability Sample
Enrollment: 479 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Prevalence of metabolic syndrome at week 13 | 13 weeks from first visit
  Change in prevalence of metabolic syndrome from baseline at week 13
Prevalence of metabolic syndrome at week 26 | 26 weeks from first visit
  Change in prevalence of metabolic syndrome from baseline at week 26
Prevalence of metabolic syndrome at week 39 | 39 weeks from first visit
  Change in prevalence of metabolic syndrome from baseline at week 39
Prevalence of metabolic syndrome at week 52 | 52 weeks from first visit
  Change in prevalence of metabolic syndrome from baseline at week 52

SECONDARY OUTCOMES:
Components of metabolic syndrome at week 13 - change in waist circumference (cm) | 13 weeks from first visit
  Baseline waist circumference data were compared with week 13 waist circumference data. Waist circumference was measured at the narrowest point of hip area or the midpoint between the lower costal (10th rib) border and the iliac crest (upper hip bone). Waist circumference data were collected in inches, and converted to cm according to the journal's requirements.
Components of metabolic syndrome at week 26 - change in waist circumference (cm) | 26 weeks from first visit
  Baseline waist circumference data were compared with week 26 waist circumference data. Waist circumference was measured at the narrowest point of hip area or the midpoint between the lower costal (10th rib) border and the iliac crest (upper hip bone). Waist circumference data were collected in inches, and converted to cm according to the journal's requirements.
Components of metabolic syndrome at week 39 - change in waist circumference (cm) | 39 weeks from first visit
  Baseline waist circumference data were compared with week 39 waist circumference data. Waist circumference was measured at the narrowest point of hip area or the midpoint between the lower costal (10th rib) border and the iliac crest (upper hip bone). Waist circumference data were collected in inches, and converted to cm according to the journal's requirements.
Components of metabolic syndrome at week 52 - change in waist circumference (cm) | 52 weeks from first visit
  Baseline waist circumference data were compared with week 52 waist circumference data. Waist circumference was measured at the narrowest point of hip area or the midpoint between the lower costal (10th rib) border and the iliac crest (upper hip bone). Waist circumference data were collected in inches, and converted to cm according to the journal's requirements.
Components of metabolic syndrome at week 13 - change in blood pressure (mmHg) | 13 weeks from first visit
  Change in blood pressure between baseline and week 13. Both blood pressures (systolic and diastolic) were assessed during the study.
Components of metabolic syndrome at week 26 - change in blood pressure (mmHg) | 26 weeks from first visit
  Change in blood pressure between baseline and week 26. Both blood pressures (systolic and diastolic) were assessed during the study.
Components of metabolic syndrome at week 39 - change in blood pressure (mmHg) | 39 weeks from first visit
  Change in blood pressure between baseline and week 39. Both blood pressures (systolic and diastolic) were assessed during the study.
Components of metabolic syndrome at week 52 - change in blood pressure (mmHg) | 52 weeks from first visit
  Change in blood pressure between baseline and week 52. Both blood pressures (systolic and diastolic) were assessed during the study.
Components of metabolic syndrome at week 13 - change in triglycerides (mmol/L) | 13 weeks from first visit
  Baseline triglycerides data were compared with week 13 triglycerides data. Mean change from baseline was measured.Triglycerides data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 26 - change in triglycerides (mmol/L) | 26 weeks from first visit
  Baseline triglycerides data were compared with week 26 triglycerides data. Mean change from baseline was measured.Triglycerides data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 39 - change in triglycerides (mmol/L) | 39 weeks from first visit
  Baseline triglycerides data were compared with week 39 triglycerides data. Mean change from baseline was measured.Triglycerides data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 52 - change in triglycerides (mmol/L) | 52 weeks from first visit
  Baseline triglycerides data were compared with week 52 triglycerides data. Mean change from baseline was measured.Triglycerides data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 13 - change in blood plasma glucose (mmol/L) | 13 weeks from first visit
  Baseline blood plasma glucose data were compared with week 13 blood plasma glucose data. Mean change from baseline was measured. Blood plasma glucose data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 26 - change in blood plasma glucose (mmol/L) | 26 weeks from first visit
  Baseline blood plasma glucose data were compared with week 26 blood plasma glucose data. Mean change from baseline was measured.Blood plasma glucose data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 39 - change in blood plasma glucose (mmol/L) | 39 weeks from first visit
  Baseline blood plasma glucose data were compared with week 39 blood plasma glucose data. Mean change from baseline was measured.Blood plasma glucose data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 52 - change in blood plasma glucose (mmol/L) | 52 weeks from first visit
  Baseline blood plasma glucose data were compared with week 52 blood plasma glucose data. Mean change from baseline was measured.Blood plasma glucose data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 13 - change in high density lipoproteins (HDL, mmol/L) | 13 weeks from first visit
  Baseline HDL data were compared with week 13 HDL data. Mean change from baseline was measured.HDL data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 26 - change in high density lipoproteins (HDL, mmol/L) | 26 weeks from first visit
  Baseline HDL data were compared with week 26 HDL data. Mean change from baseline was measured.HDL data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 39 - change in high density lipoproteins (HDL, mmol/L). | 39 weeks from first visit
  Baseline HDL data were compared with week 39 HDL data. Mean change from baseline was measured.HDL data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.
Components of metabolic syndrome at week 52 - change in high density lipoproteins (HDL, mmol/L). | 52 weeks from first visit
  Baseline HDL data were compared with week 52 HDL data. Mean change from baseline was measured.HDL data were collected in mg/dl units, and converted to mmol/L according to the journal's requirements.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Guzman M, Zbella E, Alvarez SS, Nguyen JL, Imperial E, Troncale FJ, Holub C, Mallhi AK, VanWyk S. Effect of an intensive lifestyle intervention on the prevalence of metabolic syndrome and its components among overweight and obese adults. J Public Health (Oxf). 2020 Nov 23;42(4):828-838. doi: 10.1093/pubmed/fdz170. PMID 31840755